CLINICAL TRIAL: NCT02254408
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Multi-Center Study Evaluating Antiviral Effects, Pharmacokinetics, Safety, and Tolerability of GS-5806 in Hematopoietic Cell Transplant (HCT) Recipients With Respiratory Syncytial Virus (RSV) Infection of the Upper Respiratory Tract
Brief Title: Presatovir in Hematopoietic Cell Transplant Recipients With Respiratory Syncytial Virus Infection of the Upper Respiratory Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-218-0108; 2014-002474-36 (EudraCT Number)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Respiratory Syncytial Virus
Keywords: Respiratory Syncytial Virus (RSV); Antiviral; Hematopoietic Cell Transplant (HCT); Upper respiratory tract infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — presatovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Presatovir (Experimental): Participants will receive presatovir on Days 1, 5, 9, 13, and 17, with follow-up visits through Day 28, and may continue in an optional extended monitoring phase with visits through Day 56.
  Interventions: Drug: Presatovir
- Placebo (Placebo Comparator): Participants will receive placebo on Days 1, 5, 9, 13, and 17, with follow-up visits through Day 28, and may continue in an optional extended monitoring phase with visits through Day 56.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Presatovir — Presatovir 200 mg (4 × 50 mg tablets) administered orally or via nasogastric (NG) tube
  Other Names: GS-5806
  Arms: Presatovir
Drug: Placebo — Tablets administered orally or via nasogastric tube
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of presatovir on respiratory syncytial virus (RSV) viral load in autologous or allogeneic hematopoietic cell transplant (HCT) recipients with an acute RSV upper respiratory tract infection (URTI), the effect of presatovir on development of lower respiratory tract complication, being free of any supplemental oxygen progression to respiratory failure, and pharmacokinetics (PK), safety, and tolerability of presatovir.

ELIGIBILITY:
Inclusion Criteria:

* Received an autologous or allogeneic HCT using any conditioning regimen
* Documented to be RSV-positive as determined by local testing (eg, polymerase chain reaction, direct fluorescence antibody, respiratory viral panel assay, or culture) using an upper respiratory tract sample collected ≤ 6 days prior to Day 1
* New onset of at least 1 of the following respiratory symptoms for ≤ 7 days prior to Day 1: nasal congestion, runny nose, cough, or sore throat, or worsening of one of these chronic (associated with a previously existing diagnosis, eg, chronic rhinorrhea, seasonal allergies, chronic lung disease) respiratory symptoms ≤ 7 days prior to Day 1
* No evidence of new abnormalities consistent with lower respiratory tract infection (LRTI) on a chest X-ray relative to the most recent chest X-ray, as determined by the local radiologist. If a chest X-ray is not available or was not obtained during standard care < 48 hours prior to screening, a chest X-ray must be obtained for screening
* O2 saturation ≥ 92% on room air
* An informed consent document signed and dated by the participant or a legal guardian of the participant and the investigator or his/her designee
* A negative urine or serum pregnancy test is required for female participants (unless surgically sterile or greater than two years post-menopausal)
* Male and female participants of childbearing potential must agree to contraceptive requirements as described in the study protocol
* Willingness to complete necessary study procedures and have available a working telephone or email

Exclusion Criteria:

Related to concomitant or previous medication use:

* Use of non-marketed (according to region) investigational agents within 30 days, OR use of any monoclonal anti-RSV antibodies within 4 months or 5 half-lives of screening, whichever is longer, OR use of any investigational RSV vaccines after HCT

Related to medical history:

* Pregnant, breastfeeding, or lactating females
* Unable to tolerate nasal sampling required for this study, as determined by the investigator
* Known history of HIV/AIDS with a CD4 count <200 cells/μL within the last month
* History of drug and/or alcohol abuse that, in the opinion of the investigator, may prevent adherence to study activities

Related to medical condition at screening:

* Documented to be positive for other respiratory viruses (limited to influenza, parainfluenza, human rhinovirus, adenovirus, or human metapneumovirus, or coronavirus) within 7 days prior to the screening visit, as determined by local testing (additional testing is not required)
* Clinically significant bacteremia or fungemia within 7 days prior to screening that has not been adequately treated, as determined by the investigator
* Clinically significant bacterial, fungal, or viral pneumonia within 2 weeks prior to screening that has not been adequately treated, as determined by the investigator
* Excessive nausea/vomiting at screening, as determined by the investigator, or an inability to swallow pills that precludes oral administration of the investigational medical product (for participants without an nasogastric tube in place)
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial or would interfere with the evaluation of the trial endpoints

Related to laboratory results:

* Creatinine clearance < 30 mL/min (calculated using the Cockcroft-Gault method)
* Clinically significant aspartate aminotransferase/alanine aminotransferase, as determined by the investigator
* Clinically significant total bilirubin, as determined by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (68):
- United States (27):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope, Duarte, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - NorthSide Medical Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - John Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Cancer Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
  - New York Presbyterian Hospital Cornell Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - University Hospital Case Medical, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute (SCRI), San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchison Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston
  - Royal Melbourne Hospital, Melbourne
- Brazil (7):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Fundacao Faculdade Regional Medicina de Sao Jose do Rio Preto, São Paulo
  - Fundação Antonio Prudente - Hospital do Câncer AC Camargo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital Santa Marcelina, São Paulo
  - Hospital Universitario USP, São Paulo
  - Instituto Brasileiro de Controle do Câncer-IBCC, São Paulo
- Canada (2):
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Tom Baker Cancer Centre, Calgary
- France (4):
  - CHU de Bordeaux, Bordeaux
  - Hopital Saint-Louis, APHP, Paris
  - Hopital Foch, Suresnes
  - Institut Universitaire du Cancer Oncopole, Toulouse
- Universitatsklinikum Wurzburg, Würzburg, Germany
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (2):
  - VUmc cancer center, Amsterdam
  - Erasmus Medical Center (Rotterdam), Rotterdam
- Singapore (2):
  - Singapore General Hospital, Singapore
  - UMC National University Health System, Singapore
- South Korea (5):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Hospital universitario Virgen del Rocio, Seville, Spain
- Karolinska Institutet, Stockholm, Sweden
- University Clinic Basel, Basel, Switzerland
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-LinKou Branch, Taoyuan District
- United Kingdom (2):
  - Leeds Teaching Hospitals Trust, Leeds
  - King's College Hospital, London

REFERENCES:
- [Derived] Chemaly RF, Dadwal SS, Bergeron A, Ljungman P, Kim YJ, Cheng GS, Pipavath SN, Limaye AP, Blanchard E, Winston DJ, Stiff PJ, Zuckerman T, Lachance S, Rahav G, Small CB, Mullane KM, Patron RL, Lee DG, Hirsch HH, Waghmare A, McKevitt M, Jordan R, Guo Y, German P, Porter DP, Gossage DL, Watkins TR, Marty FM, Chien JW, Boeckh M. A Phase 2, Randomized, Double-blind, Placebo-Controlled Trial of Presatovir for the Treatment of Respiratory Syncytial Virus Upper Respiratory Tract Infection in Hematopoietic-Cell Transplant Recipients. Clin Infect Dis. 2020 Dec 31;71(11):2777-2786. doi: 10.1093/cid/ciz1166. PMID 31793991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in North America, Europe, Australia and Asia. The first participant was screened on 23 January 2015 and the last study visit occurred on 14 July 2017.
Pre-assignment Details: 213 participants were screened.
Groups:
- Presatovir: Presatovir 200 mg (4 x 50 mg tablets) administered as a single dose, orally or via nasogastric (NG) tube on Days 1, 5, 9, 13, and 17
- Placebo: Placebo administered orally or via NG tube on Days 1, 5, 9, 13, and 17
Period: Overall Study
Arm/Group | Presatovir | Placebo
Started | 96 | 93
Completed | 88 | 83
Not Completed | 8 | 10
Not completed — Randomized But Not Treated | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Death | 2 | 3
Not completed — Investigator's Discretion | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study medication
Groups:
- Presatovir: Presatovir 200 mg (4 x 50 mg tablets) administered as a single dose, orally or via NG tube on Days 1, 5, 9, 13, and 17
- Total: Total of all reporting groups
Arm/Group | Presatovir | Placebo | Total
Number analyzed (Participants) | 95 | 90 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (12.21) | 51.4 (14.58) | 51.8 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 35 | 75
  Male | 55 | 55 | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 9 | 22
  Black or African American | 6 | 3 | 9
  White | 66 | 70 | 136
  Other | 2 | 0 | 2
  Not Permitted | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 81 | 75 | 156
  Not Permitted | 6 | 9 | 15
Region of Enrollment [Number; unit: participants] — All Randomized Analysis Set: all participants randomized in the study.
  participants
    Singapore | 3 | 2 | 5
    United States | 58 | 55 | 116
    United Kingdom | 3 | 2 | 5
    Switzerland | 0 | 1 | 1
    Canada | 3 | 5 | 8
    South Korea | 5 | 1 | 6
    Israel | 10 | 11 | 21
    Australia | 6 | 3 | 9
    France | 7 | 10 | 18
Nasal Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] — Population: Participants in the Safety Analysis Set with available data were analyzed.
  log10 copies/mL
    number analyzed (Participants) | 95 | 88 | 183
    (all) | 6.31 (1.899) | 6.51 (1.437) | 6.41 (1.691)

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Average Change in Nasal Respiratory Syncytial Virus (RSV ) Viral Load From Baseline (Day 1) to Day 9
Description: The time-weighted average change, often referred to as the DAVG, provides the average viral burden change from baseline. The mean values presented were calculated using the ANCOVA model and are adjusted for baseline value and stratification factor.
Time Frame: Baseline; Day 9
Population: Full Analysis Set: participants who received at least 1 full dose of study drug and had an RSV viral load greater than or equal to the lower limit of quantification of the quantitative real-time polymerase chain reaction (RT-qPCR) assay in the Day 1 nasal sample, as determined by RT-qPCR.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 89 | 87
log10 copies/mL | -1.26 (0.964) | -0.91 (1.145)
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.040, ANCOVA; Treatment Difference = -0.33, 95% CI 2-sided [-0.64 to -0.02]

2. Primary Outcome: Percentage of Participants Who Developed a Lower Respiratory Tract Complication
Description: A Lower Respiratory Tract Complication (LRTC) was defined as one of the below as determined by the adjudication committee:
  * Primary RSV lower respiratory tract infection (LRTI)
  * Secondary bacterial LRTI
  * LRTI due to unusual pathogens
  * Lower respiratory tract complication of unknown etiology
Time Frame: Up to Day 28
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 89 | 87
percentage of participants | 11.2 [5.5 to 19.7] | 19.5 [11.8 to 29.4]
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.11, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.22 to 1.18]
Statistical Analysis 2: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.15, Fisher Exact

3. Secondary Outcome: Percentage of Participants Who Developed Respiratory Failure (of Any Cause) Requiring Mechanical Ventilation (Invasive or Noninvasive) or All-cause Mortality
Description: Participants were considered to have an event if either condition is met:
  * Participant develops a respiratory failure (of any cause) requiring mechanical ventilation (invasive or noninvasive) or;
  * Participant dies prior to or on Day 28
Time Frame: Up to Day 28
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 89 | 87
percentage of participants | 5.6 [1.8 to 12.6] | 5.7 [1.9 to 12.9]
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.98, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.28 to 3.63]
Statistical Analysis 2: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 1.00, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Safety Analysis Set
Arm/Group | Presatovir | Placebo
All-Cause Mortality (participants affected / at risk) | 2/95 | 4/90
Serious Adverse Events (participants affected / at risk) | 18/95 | 23/90
Other Adverse Events (participants affected / at risk) | 49/95 | 47/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Presatovir (N=95) | Placebo (N=90)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Food allergy (Immune system disorders) | 0 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2 | 0
Clostridial sepsis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 6
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 3
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Presatovir (N=95) | Placebo (N=90)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 5
Neutropenia (Blood and lymphatic system disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 15 | 14
Nausea (Gastrointestinal disorders) | 13 | 10
Vomiting (Gastrointestinal disorders) | 10 | 12
Asthenia (General disorders) | 3 | 7
Pyrexia (General disorders) | 10 | 9
Decreased appetite (Metabolism and nutrition disorders) | 7 | 6
Dizziness (Nervous system disorders) | 7 | 3
Headache (Nervous system disorders) | 5 | 7
Acute kidney injury (Renal and urinary disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (8):
  • Study Protocol: Original (2014-05-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT02254408/Prot_000.pdf
  • Study Protocol: Amendment 1 (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT02254408/Prot_001.pdf
  • Study Protocol: Amendment 2 (2014-09-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT02254408/Prot_002.pdf
  • Study Protocol: Amendment 3 (2014-10-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT02254408/Prot_003.pdf
  • Study Protocol: Amendment 5 (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT02254408/Prot_004.pdf
  • Study Protocol: Amendment 6 (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT02254408/Prot_005.pdf
  • Study Protocol: Amendment 7 (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02254408/Prot_006.pdf
  • Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02254408/SAP_007.pdf